CLINICAL TRIAL: NCT05137873
Title: Measurement of the Prevalence of Sensory Integration Disorders in Babies Having Heart Disease Surgery for Transposition of the Great Vessels Before 6 Months of Age
Acronym: SENSOCOEUR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other); Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211266; 2021-A02294-37 (Other: ID-RCB)
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Great Vessels Transposition Surgery
Keywords: sensory integration disorders; great vessels transposition surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery before 6 months of age: Babies with heart disease surgery, great vessels transposition surgery type before 6 months of age
  Interventions: Other: Dunn-2 infant Sensory Profile (PS2-N)

INTERVENTIONS:
Other: Dunn-2 infant Sensory Profile (PS2-N) — The Dunn-2 infant Sensory Profile evaluates the child's sensory integration process

SUMMARY:
The purpose of this study is to mesure the prevalence of severe sensory integration disorders in babies after one week of their heart surgery.

DETAILED DESCRIPTION:
Baby's development takes its roots in sensorimotricity. Baby coordinates different senses (visual, auditory, tactile, taste, vestibular) to understand the space around him and to implement voluntary motor strategies. These sensory links also allow him to invest hisoral zone and consolidate his oral feeding. Another good sensory integration is necessary for a child to develop harmoniously on motor and psychic levels. In 2018 the study of L. Dagenais revealed a gap in posturomotor development on babies operated on for isolated congenital heart disease. However nobody assess sensory disorders in these babies. With this study the investigators wish to clarify the sensory impact in this situation.

ELIGIBILITY:
Inclusion Criteria:

* Infant born at term (over 37 weeks)
* With heart disease, of the transposition of the great vessels type, whether or not associated with an interventricular communication
* Having a cranial perimeter in the norm at birth: between 32 and 37 cm.
* Surgery scheduled before the age of 6 months
* No opposition from parents

Exclusion Criteria:

* Other disease or malformation
* Parents who do not speak French

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies with heart disease surgery, great vessels transposition surgery type before 6 months of age
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The Dunn-2 infant Sensory Profile Score one week after surgery | 1 week after surgery
  The Dunn-2 infant Sensory Profile evaluates a child's sensory integration process. PS2-N has 25 variables rated from 0 to 5.
  The sum of these variables is the total raw score:
  0 to 30: much less than others 31 to 40: less than the others 41 to 61 : Like the majority 62 to 71: more than the others 72 to 125 : much less than the others

SECONDARY OUTCOMES:
The Dunn-2 infant Sensory Profile Score one month after surgery | 1 month after surgery
  The Dunn-2 infant Sensory Profile evaluates a child's sensory integration process
The Dunn-2 infant Sensory Profile Score 6 months after surgery | 6 months after surgery
  The Dunn-2 infant Sensory Profile evaluates a child's sensory integration process
Eating disorders one week after surgery | 1 week after surgery
  Eating disorders are assessed by the Montréal Children's Hospital (HME) feeding scale. HME feeding scale has 14 variables rated from 1 to 7.
  A score above 45 identifies feeding problems
Eating disorders one month after surgery | 1 month after surgery
  Eating disorders are assessed by the HME feeding scale
Eating disorders 6 months after surgery | 6 months after surgery
  Eating disorders are assessed by the HME feeding scale
Implementation of functional rehabilitation 1 month after surgery | 1 month after surgery
  Collection of physiotherapy and psychomotricity needs
Implementation of functional rehabilitation 6 months after surgery | 6 months after surgery
  Collection of physiotherapy and psychomotricity needs

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Abadie, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker - Enfants malades hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dagenais L, Materassi M, Desnous B, Vinay MC, Doussau A, Sabeh P, Prud'homme J, BSc KG, Lenoir M, Charron MA, Nuyt AM, Poirier N, Beaulieu-Genest L, Carmant L, Birca A. Superior Performance in Prone in Infants With Congenital Heart Disease Predicts an Earlier Onset of Walking. J Child Neurol. 2018 Dec;33(14):894-900. doi: 10.1177/0883073818798194. Epub 2018 Sep 18. PMID 30226082
- [Background] Abadie V. [Apparently isolated feeding behavior troubles in infant]. Arch Pediatr. 2008 Jun;15(5):837-9. doi: 10.1016/S0929-693X(08)71932-8. No abstract available. French. PMID 18582771
- [Background] Dunn W, Westman K. The sensory profile: the performance of a national sample of children without disabilities. Am J Occup Ther. 1997 Jan;51(1):25-34. doi: 10.5014/ajot.51.1.25. PMID 8978860
- [Background] Ramsay M, Martel C, Porporino M, Zygmuntowicz C. The Montreal Children's Hospital Feeding Scale: A brief bilingual screening tool for identifying feeding problems. Paediatr Child Health. 2011 Mar;16(3):147-e17. doi: 10.1093/pch/16.3.147. PMID 22379377